CLINICAL TRIAL: NCT05682651
Title: Etiological Investigation of 'Post-Intubation Tracheal Stenosis' Cases Requiring Intervention: 2-year Case Review
Brief Title: Relationship Between Post-Intubation Tracheal Stenosis and Covid-19
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nilgün Zengin, Principal İnvestigator, Ankara City Hospital Bilkent
Other Study IDs: E.Kurul-E1-22-3142
Record Dates: First submitted 2023-01-07; First posted 2023-01-12 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Tracheal Stenosis; COVID-19; Post-Intubation Subglottic Stenosis; Intensive Care Unit
MeSH Terms: conditions — Tracheal Stenosis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tracheal Stenosis with Covid-19: Patients' age, gender, American Society of Anesthesiologists (ASA) classification, comorbidities, etiologic cause, intubation time, type of surgery, length of hospital stay, and morbidity/mortality information will be recorded.
  Interventions: Procedure: tracheal stenosis follow-up file
- Tracheal Stenosis with Non-Covid-19: Patients' age, gender, American Society of Anesthesiologists (ASA) classification, comorbidities, etiologic cause, intubation time, type of surgery, length of hospital stay, and morbidity/mortality information will be recorded.
  Interventions: Procedure: tracheal stenosis follow-up file

INTERVENTIONS:
Procedure: tracheal stenosis follow-up file — Patients' age, gender, American Society of Anesthesiologists (ASA) classification, comorbidities, etiologic cause, intubation time, type of surgery, length of hospital stay, and morbidity/mortality information will be recorded.

SUMMARY:
Tracheal stenosis (TS) is a serious complication that occurs in approximately 6-22% of patients due to prolonged endotracheal intubation. Cuff hyperinflation of the endotracheal tube, use of large tubes, advanced age, female gender, smoking, obesity, and diabetes are risk factors for TS. The most common and serious complication in COVID-19 patients is acute respiratory distress syndrome (ARDS), which requires oxygen and ventilation treatments. In the literature, it is reported that 9.8-15.2% of patients need invasive mechanical ventilation (IMV). The concern of aerosol formation and prone position applications that emerged with the coronavirus pandemic caused delays in tracheostomy decisions and the use of uncontrolled high cuff pressures, paving the way for TS. The capillary perfusion pressure of the tracheal mucosa ranges from 20 to 30 mmHg. A cuff pressure of the endotracheal tube above 30 mmHg causes mucosal ischemia. Cartilage inflammation due to ischemic injury may be partial or full thickness. Depending on the degree of inflammation in the affected tracheal segments, stenosis and even perforation may develop.

It is aimed to determine the etiological causes, to determine how much of the total TS cases covid-related TS constitutes, to examine the treatments and patient results in covid/non-covid TS.

This study will contribute to the measures that can be taken during and after the care process in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years

Exclusion Criteria:

* Patients undergoing surgical procedures for malignancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age and without a history of malignancy who developed post-intubation tracheal stenosis are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-05-28 (Actual)

PRIMARY OUTCOMES:
Intubation time | Up to 3 months
  Duration of intubation of patients (in days)
Morbidity/mortality | Up to 2 months
  Morbidity/mortality status of the patients within 3 months
Length of hospital stay | Up to 3 months
  The hospital stay of the patients will be recorded (in days)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Çankaya, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No